CLINICAL TRIAL: NCT04056728
Title: A Prospective, Open-label, Interventional Phase IV Study to Assess the Safety of EupentaTM Inj. {Fully Liquid Pentavalent Vaccine, Adsorbed Diphtheria-Tetanus-whole-cell Pertussis-Hepatitis B (rDNA [Recombinant-deoxyribonucleic Acid])-Haemophilus Influenzae Type b Conjugate Vaccine}
Brief Title: A Phase IV Study to Assess the Safety of EupentaTM Inj
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LG-VPCL005
Record Dates: First submitted 2019-08-01; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis B; Diphtheria; Haemophilus Influenzae Type B Infection; Tetanus; Pertussis
MeSH Terms: conditions — Hepatitis B; Diphtheria; Haemophilus Infections; Tetanus; Whooping Cough

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eupenta Inj. (Experimental)
  Interventions: Biological: Eupenta Inj.

INTERVENTIONS:
Biological: Eupenta Inj. — fully liquid pentavalent vaccine, Adsorbed Diphtheria-Tetanus-whole-cell Pertussis-Hepatitis B (rDNA [recombinant-deoxyribonucleic acid])-Haemophilus influenzae type b conjugate vaccine single dose 0.5 mL/vial The vaccine is given at 6, 10 and 14 weeks of age in infants.

SUMMARY:
A prospective, open-label, interventional phase IV study to assess the safety of EupentaTM Inj.{fully liquid pentavalent vaccine, Adsorbed Diphtheria-Tetanus-whole-cell Pertussis-Hepatitis B (rDNA [recombinant-deoxyribonucleic acid])-Haemophilus influenzae type b conjugate vaccine}

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the parents or legally acceptable representatives (LARs) of the subject who have been informed of the purpose, method, effects, etc., of the study
2. A male or female 6 to 8 weeks of age, inclusive, at the time of the first vaccination
3. In good health as determined by medical history, physical examination, and judgment by the Investigator
4. Body weight 3.2 kg and over at the time of screening
5. Subjects for whom the Investigator believed that their parent(s)/LAR(s) could comply with the requirements of the protocol (e.g., completion of the Subject Diary Cards, return for site visits)

Exclusion Criteria:

1. Past or present medical history of known or suspected diphtheria, tetanus, pertussis, polio, HB and/or Hib diseases
2. Any history of allergy to any of the components or excipients of EupentaTM Inj., including aluminum hydroxide, sodium hydrogen phosphate heptahydrate, monobasic sodium phosphate dihydrate, polysorbate and thimerosal
3. Any medical condition which can compromise the infant's safety, as per Investigator's discretion
4. History of seizures or abnormal cerebral signs in the newborn period or other serious neurological abnormality
5. History of bleeding tendencies
6. Household contact and/or intimate exposure with a confirmed case of diphtheria, pertussis, HB, polio and/or Hib diseases within in 30 days prior to screening
7. History of fever ≥ 38°C/ 100.4°F within 3 days prior to screening and/or intake of anti-pyretic/analgesic medication. Subjects who meet this criterion will be rescreened to check the temperature after the temporary condition has resolved and if they are within the window period for age of first vaccination at the time of re-scheduled visit
8. History of previous diphtheria-tetanus-pertussis (DTP), and/or Hib vaccination doses
9. History of previous or concurrent vaccinations other than Bacillus Calmette-Guérin (BCG), HB vaccination at birth, Polio, Rotavirus and Pneumococcal vaccines
10. Known or suspected immune disorders, or, received immunosuppressive therapy
11. Participation 30 days prior to screening in the study or simultaneously in another study and/or received any investigational product

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2019-09-23 (Estimated); Primary Completion 2020-10-12 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of any immediate reactions reported from the study after EupentaTM Inj. Vaccination | first 30 minutes after each study vaccination
Incidence of solicited local and systemic adverse events (AEs) | baseline(pre-vaccination) up to 7 days after each vaccination
Incidence of any unsolicited AEs during the entire study | through study completion, an average of 1 year
Incidence of SAEs during the entire study period | through study completion, an average of 1 year